CLINICAL TRIAL: NCT02085265
Title: The SARTAN-AD Trial: A Randomized, Open Label, Proof of Concept Study of Telmisartan vs. Perindopril in Mild-Moderate Alzheimer's Disease Patients
Brief Title: Telmisartan vs. Perindopril in Mild-Moderate Alzheimer's Disease Patients
Acronym: SARTAN-AD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Weston Brain Institute (Other)
Responsible Party: Principal Investigator, Dr. Sandra E Black, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 148-2013
Record Dates: First submitted 2013-11-29; First posted 2014-03-12 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Perindopril; Telmisartan; Brain atrophy
MeSH Terms: conditions — Alzheimer Disease | interventions — Perindopril; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Telmisartan (Experimental): Telmisartan 40 mg or 80 mg/day (depending on age and tolerability)
  Interventions: Drug: Telmisartan
- Perindopril (Active Comparator): Perindopril 2 mg, 4 mg or 8 mg/day (depending on kidney function and tolerability)
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: Perindopril — Perindopril 2 mg, 4 mg or 8 mg/day (depending on kidney function and tolerability)
  Other Names: Coversyl
  Arms: Perindopril
Drug: Telmisartan — Telmisartan 40 mg or 80 mg/day (depending on age and tolerability)
  Other Names: Micardis
  Arms: Telmisartan

SUMMARY:
To conduct a proof of concept study in patients with mild to moderate Alzheimer's Disease in order to determine if there is less global brain atrophy over one year, as measured by ventricular enlargement as a primary outcome measure, when patients are randomized to treatment with an angiotensin receptor blocker (ARB) compared to an angiotensin converting enzyme inhibitor (ACEI).

DETAILED DESCRIPTION:
This study uses a simple validated measure of brain atrophy as a surrogate marker in a repurposing effort that could recast an antihypertensive medication as a cognitive enhancer/neuroprotective agent and possibly as a drug of choice for Alzheimer patients and patients at risk for AD. If the proof of concept result is positive, a larger study would be warranted with potential practice-changing impact.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of Probable AD dementia or Possible AD dementia due to concomitant cerebrovascular disease (as permitted by the study exclusion criteria), using the 2011 McKhann criteria.
2. Previous brain MRI or CT scan to rule out exclusionary pathology, and absence of stepwise decline since the previous scan.
3. Age 50 years or older
4. Standardized Mini Mental State Examination (SMMSE) score of 16-27 at screening visit
5. Sufficient hearing and vision to participate in testing as per investigator's judgement
6. Sufficient fluency in English to understand instructions and to be able to complete SMMSE
7. A study partner who in the opinion of the study investigator has regular interaction with the participant, can be present for study visits, can provide a collateral history and can ensure compliance with study procedures
8. HbA1C <8.5%. Patients with stable type II diabetes are eligible for the study if there have been no severe hypoglycemic events requiring third party intervention (e.g. emergency department visit) for 6 months prior to randomization
9. Patients on cholinesterase inhibitors or memantine, medications for vascular risk factors (e.g., hypertension, cholesterol, diabetes), or on psychotropic medications must be on a stable dose for 30 days prior to randomization.

Exclusion criteria

1. Intolerance, or any contraindications, to study medications
2. Average SBP <110mmHg or average DBP <60 mmHg during screening
3. Familial autosomal dominant form of Alzheimer's disease
4. Creatinine clearance less than or equal to 30ml/min
5. Serum potassium > 5.5 mEq/L
6. ALT 3x > the upper limit of normal (ULN)
7. History of angioedema
8. Co-morbid acute or chronic conditions (including type I diabetes mellitus, other neurological conditions such as Parkinson's disease, psychiatric disorders, and severe or unstable medical conditions) that could confound assessments or would, in the judgment of the investigator, make the subject inappropriate for entry into this study
9. Any of the following findings on previous CT/MRI or on screening MRI:

   Exclusionary Finding: Malignant tumour Brain Location: Anywhere Size: Any Exclusionary Number: Any

   Exclusionary Finding: Tumour with significant mass effect Brain Location: Anywhere Size: Sufficient for mass effect Exclusionary Number: Any

   Exclusionary Finding: Vascular malformations Brain Location: Anywhere Size: Any Exclusionary Number: Any

   Exclusionary Finding: Subdural hematoma Brain Location: Anywhere Size: Any Exclusionary Number: Any

   Exclusionary Finding: Intracerebral hemorrhage Brain Location: Anywhere Size: Any Exclusionary Number: Any

   Exclusionary Finding: Cerebral microbleeds, Brain Location: Anywhere Size: Any Exclusionary Number: more than 5

   Exclusionary Finding: Superficial siderosis (SS) Brain Location: Cortex Size: Any Exclusionary Number: >1 instance of focal SS

   Exclusionary Finding: Ischemic infarct Brain Location: Cortex Size: >1.5 cm in diameter Exclusionary Number: Any

   Exclusionary Finding: Ischemic infarct Brain Location: Cortex Size: ≤1.5 cm in diameter Exclusionary Number: more than 1

   Exclusionary Finding: Fazekas score 3 with white matter hyperintensity band along the lateral surface of the ventricles >0.5 cm in width

   Exclusionary Finding: Ischemic infarct Brain Location: White matter Size: >1.5 cm in diameter Exclusionary Number: Any

   Exclusionary Finding: Ischemic infarct Brain Location: White matter Size: 1.0-1.5 cm in diameter Exclusionary Number: More than 2

   Exclusionary Finding: Ischemic infarct Brain Location: Basal ganglia Size: >1.0 cm in diameter Exclusionary Number: Any

   Exclusionary Finding: Ischemic infarct Brain Location: Basal ganglia and white matter Size: ≤1.0 cm in diameter Exclusionary Number: More than 4

   Exclusionary Finding: Strategic infarct Brain Location: Thalamus Size: Any Exclusionary Number: Any

   Exclusionary Finding: Strategic infarct Brain Location: Hippocampus, Size: Any Exclusionary Number: Any
10. Inability to perform the study procedures, including claustrophobia or contraindications for MRI
11. Currently on or has taken an angiotensin receptor blocker within 12 months of randomization visit
12. Resides in a nursing home (participants who reside in retirement homes may be included if they have a study partner who meets inclusion criterion #8)
13. Current major depression by clinical history or score greater than 18 on the Cornell Scale for Depression in Dementia
14. Documented potential cardiac source of brain infarction such as mechanical valve or atrial fibrillation that is untreated or treated with warfarin or an antiplatelet agent; atrial fibrillation treated with a novel oral anticoagulant is permitted, as is a history of remote, transient atrial fibrillation that has not recurred

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Ventricular enlargement | 12 months
  Change in ventricular size, on 3D T1 MR imaging, after 12 months of treatment
Safety - Blood pressure | 12 months
  Change in blood pressure (BP) measurements after 12 months of treatment.
Safety - Vital signs | 12 months
  Change in vital sign (heart rate, pulse) measurements after 12 months of treatment.
Safety - Electrolytes | 12 months
  Change in electrolyte measurements (Na, K) after 12 months of treatment.
Safety - Adverse Events | 12 months
  Adverse events and serious adverse events over 12 months of treatment.

SECONDARY OUTCOMES:
Hippocampal volume | 12 months
  Change in hippocampal volume measurements after 12 months of treatment
Grey/White matter volume | 12 months
  Volume of grey and white matter in the cingulate, parietotemporal and dorsolateral frontal regions after 12 months of treatment
Cognitive and functional measures | 6 and 12 months
  Determine comparative efficacy of perindopril vs. telmisartan on cognitive and functional measures and on other structural brain imaging measures in this participant population

OTHER OUTCOMES:
Neuropsychiatric Measures | 6 & 12 months
  Assess the comparative treatment responsiveness of neuropsychiatric measures and obtain pilot data
Treatment responsiveness of Diffusion Tensor Imaging (DTI) | 12 months
  Assess the comparative treatment responsiveness of Diffusion Tensor Imaging (DTI) and obtain pilot data
Treatment responsiveness of resting state functional MRI (rsfMRI) | 12 months
  Assess the comparative treatment responsiveness of multi-modal MRI, resting-state functional MRI (rsfMRI) and arterial spin labeling (in a subset of participants) and obtain pilot data.
Quality of Life - Caregiver burden | 12 months
  Assess the comparative response of caregiver burden after treatment using Zarit burden interview.
Quality of Life - Health-related | 12 months
  Assess health related quality of life after treatment using EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Black, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Krista Lanctot, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (10):
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - University of Lethbridge, Lethbridge, Alberta
  - UBC Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Parkwood Institute, London, Ontario
  - Centre for Memory and Aging, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario